CLINICAL TRIAL: NCT06572865
Title: Identifying Parents in Child Welfare Services Who Need Mental Health Support: Depression and Anxiety Symptoms and Associated Factors
Brief Title: Identifying Parents in Child Welfare Services Who Need Mental Health Support: Depression and Anxiety Symptoms
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Martin Forster, Principal Investigator, Karolinska Institutet
Other Study IDs: Parent symptoms CWS
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mental Illness; Depression; Anxiety
Keywords: Mental Illness; Depression; Anxiety; Parenting
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parents reported to the child welfare services: Adults who are into contact with the Swedish CWS due to a child welfare report. The adults have a parental role in relation to a child 0-17 years old (referred to as 'parents').
  Interventions: Other: Screening for depression and anxiety

INTERVENTIONS:
Other: Screening for depression and anxiety — Parents respond to questionnaires assessing depression and anxiety.

SUMMARY:
The main aim of this study is to examine the occurrence of mental health symptoms among parents referred to the Swedish child welfare services for child maltreatment and other family related risks. Additionally, to examine any variables associated with parents' levels of depression and anxiety.

Parents will respond to questionnaires administered by social workers. The level of depression and anxiety will be descriptively and statistically compared to clinical and normative samples. Additionally, statistical analyses will examine variables associated with parents' mental health symptoms.

DETAILED DESCRIPTION:
BACKGROUND:

Parental mental illness is associated with various family-related risks, including child maltreatment and children developing own psychiatric conditions. Studies indicate that parental mental illness is more prevalent in families into contact with the child welfare system due to child maltreatment or other risk conditions. However, there is a lack of studies that routinely examine the well-being of parents reported for child maltreatment. Furthermore, there is limited knowledge of whether the severity of parental symptoms varies based on the reasons for the child welfare report.

PURPOSE AND RESEARCH QUESTIONS:

The main aim of this study is to assess the occurrence of mental health symptoms among parents referred to the child welfare services (CWS) and whether any factors are associated with the level of symptoms. The research questions are:

1. Is the average level of depression and anxiety among parents reported to CWS different from that in normative and clinical populations?
2. Are parent and family characteristics, the reason for the child welfare involvement, or previous involvement with CWS associated with parents' levels of depression and anxiety?

METHODS:

This is a cross-sectional study using data collected within a feasibility study of the Collaboration-Screening-Referral model (in Swedish: Samverkan-Screening-Hänvisning - SSH) - an approach to screen parents for symptoms of mental illness using structured questionnaires, establish intra-agency collaboration, and refer to mental health services. An evaluation of the effects, feasibility and experiences of the SSH-model is presented in a separate study: "Screening to Identify Parents in Need of Mental Health Support: A Feasibility Study in Child Welfare Services". The present study presents data from the questionnaire administered to parents.

CWS agencies in Swedish municipalities will be recruited to take part in the research project. Social workers will receive training in employing screening for depression and anxiety. Then, they will administer a questionnaire measuring symptoms of depression and anxiety to parents they meet as a part of routine work. They will be encouraged to present the screening to every eligible parent they meet. When parents have responded to questionnaires, it is followed by a discussion about well-being and support needs. When relevant, the social worker provides information about what mental health support is available.

Parents' data will be anonymous. The multiple-choice questions will be restricted and phrased in a way that prevents identification. The survey will be made available in several languages.

SAMPLE SIZE CALCULATION AND ANALYSES:

Mean values from the instruments will be presented descriptively. Also, compared statistically (using t-test or ANOVA) to established cut-off values/clinical samples as well as data from parents in the general population. To take account of possible nesting effects resulting of parents from the same families responding, the alpha will conservatively be set to 0.025. At least 290 participants are needed for an 80% power (alpha = 0.025) to detect a small mean difference (d = 0.20). Additionally, multiple linear regression analyses will examine variables associated with parents' symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A parental role in relation to a child 0-17 years old (the participant does not be a guardian or biological parent, can also be, for example, a partner to a parent).
* A child welfare report has been filed for the child or the parent has reached out to the CWS themselves.

Exclusion Criteria:

* Not able to read questionnaire in any available language and interpreter not available at the social services.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents reported to the social services due to concerns of the child's well-being.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire | At inclusion, each participant will be assessed one time only.
  The Patient Health Questionnaire (PHQ-9) will be used to assess depressive symptoms, including suicidal ideation, over the last two weeks (9 questions). Items are scored 0-3, resulting in a total score of 0-27. Higher scores indicate more symptoms of depression.
The GAD-7 | At inclusion, each participant will be assessed one time only.
  The 7-item GAD-7 will measure symptoms of anxiety. Items are scored 0-3, resulting in a total score of 0-21. Higher scores indicate more symptoms of anxiety.

SECONDARY OUTCOMES:
Parents' background | At inclusion, each participant will be assessed one time only.
  Parent will respond to a few questions about their background when responding to the screening questionnaire.
Parents' contact with mental health services | At inclusion, each participant will be assessed one time only.
  In the screening questionnaire, parents will be asked whether they are currently or have previously been in contact with healthcare services for their mental health.
Characteristics of the contact with child welfare services | At inclusion, each participant will be assessed one time only.
  In the parents' questionnaires, previous contact with child welfare services will be recorded, along with the reason for the current involvement with child welfare services.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No